CLINICAL TRIAL: NCT07343596
Title: Study to Identify Biomarkers of Oral Cavity Cancer Response to Neoadjuvant Immunotherapy Prior to Definitive Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-1536; A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); Protocol Version 12/30/25 (Other: UW Madison); UW25009 (Other: UW Madison)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Oral Cavity Cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Standard of Care: Pembrolizumab (Experimental): Participants receive pembrolizumab by a needle (IV) in the arm once per standard of care (SOC)
  Interventions: Biological: Pembrolizumab; Device: Patient-Specific Culture Vessel

INTERVENTIONS:
Biological: Pembrolizumab — IV injection of pembrolizumab
Device: Patient-Specific Culture Vessel — LumeNEXT platform, which employs a 3D matrix and allows molding of blood and lymphatic vessels

SUMMARY:
The goal of this clinical trial is to study whether researchers can create a patient-specific tumor system, called a culture vessel, in a timely manner and determine if it can predict how someone will respond to a specific therapy.

Participants will:

* Undergo a research biopsy
* Take pembrolizumab per standard of care prior to surgery

DETAILED DESCRIPTION:
Immunotherapy has improved survival for selected patients with recurrent/metastatic head and neck cancer. The Keynote-689 study results published in the New Eng J Med demonstrating improved event free survival for head and neck cancer patients receiving pembrolizumab prior to surgery prompted the June 12, 2025 FDA approval of pembrolizumab as a standard of care option. However, selecting those patients most likely to benefit from this approach is challenging due to a lack of predictive biomarkers.

In this trial, the team will investigate biomarkers using single cell RNA sequencing and a patient-specific culture vessel. These models will not be used to make clinical decisions in this study. Rather, to explore whether a patient-specific culture vessel readout may be feasible to incorporate within a clinical trial workflow. If this proves feasible within an 8-week timeframe, and promising biomarkers of response are identified, this culture vessel may be worthy to study further in subsequent clinical trials.

The investigators chose 2 months as a time point because it is quicker than physicians can currently determine patient overall response (typically 4-6 months) to immunotherapy and still long enough to allow the model to be developed and tested appropriately.

Primary objective: To identify biomarkers predicting treatment response to neoadjuvant immunotherapy in oral cavity cancer

Secondary objectives:

* To correlate tumor response to immunotherapy in the patient-specific culture vessel to clinical tumor response to immunotherapy in vivo (the patient) after treatment with pembrolizumab immunotherapy.
* To determine the feasibility of utilizing the patient-specific culture vessel within a clinical trial workflow.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* Age 18 years and older at the time of registration consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 within 30 days prior to enrollment
* Suspected clinical American Joint Committee on Cancer (AJCC) 8th edition stage II-IVB (T2-T4b N0-N3) oral cavity cancer (oral tongue, floor of mouth, buccal, gingival, retromolar trigone, lip, hard palate) amenable to surgical resection. Patients will be consented prior to research biopsy.
* Primary tumor of at least 2 cm which is amenable to a 250 mm3 (e.g.10 mm x 5 mm x 5 mm) research biopsy, equivalent to one-two forceps biopsies.
* Patients may not have received prior chemotherapy or immunotherapy for the oral cavity malignancy. Patients must have completed other cancer therapies unrelated to their oral cavity cancer greater than 30 days prior to enrollment.
* Participants of childbearing potential must agree to contraception during and for 100 days after study therapy.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to treatment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for > 12 consecutive months.
* Demonstrate adequate organ function

Exclusion Criteria:

* Subjects with a diagnosed auto-immune disease (exceptions: subjects with controlled diabetes mellitus type I, thyroid disease, rheumatoid arthritis, vitiligo and alopecia areata not requiring treatment with immunosuppressants are eligible)
* Pregnant or breastfeeding
* Known additional invasive malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease free for at least three years prior to enrollment. This excludes the index oral cavity cancer.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor.
* Has received prior radiotherapy treatment or systemic anti-cancer therapy including investigational agents for the HNC under study prior to randomization/allocation.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has had previous allogeneic tissue/solid organ transplant.
* Subjects who require systemic treatment doses of corticosteroids (prednisone equivalent greater than or equal to 10 mg daily), or other immunosuppressive drugs
* Has radiographically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis as assessed by local site investigator and radiology review
* Has Grade 3-4 bleeding due to the underlying malignancy
* Subjects with known human immunodeficiency virus (HIV) infection, active or chronic hepatitis B or hepatitis C infection based on medical history. No testing for HIV, Hepatitis B, or Hepatitis C is required for enrollment. Subjects cannot be positive for HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-hepatitis B core antibody. Patients with Hepatitis B surface antigen negative and anti-hepatis B core antibody positive with undetectable HBV DNA by polymerase chain reaction may enroll.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
* Subjects who cannot provide independent, legal, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Gene Expression | up to 2 months
  Identification of pathways that are activated in samples showing substantial response versus those that do not. Gene expression changes will be evaluated through mRNA sequencing and bioinformatic analysis.
Phenotypic Changes in the Immune Microenvironment | up to 2 months
  Pathways critical for immune response will be assessed using microscopy and a custom analysis pipeline to assess changes in immune cell localization, staining and morphology that will be compared to a control condition and reported as increased or decreased compared to control. Secreted factors will be assessed in culture media using multiplex bead-based ELISA and quantification of secreted factors will be reported as a concentration (pg/ml or ng/ml) and compared to determine increase or decrease compared to control condition.
Genotypic Changes in the Immune Microenvironment | up to 2 months
  Genotypic changes will be assessed using bulk or single cell sequencing approaches. Differential gene expression between control and treatment conditions will be reported and compared between conditions. Gene enrichment pathway analysis will also be completed and compared between control and treatment conditions. For single cell sequencing analysis identified cell clusters will be compared between treatment conditions.

SECONDARY OUTCOMES:
Tumor response | 8 weeks
  Tumor response in the pathologic specimen is assessed by the area of treatment effect. This is defined as the area of tumor necrosis with associated keratinaceous debris. It will be reported as the ratio of the area of tumor effect divided by the total area of tumor.
Feasibility of implementation of a patient-specific culture vessel | 8 weeks
  Feasibility is defined as availability of patient-specific culture vessel data.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Burr, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes